CLINICAL TRIAL: NCT06635226
Title: A Randomized, Double-blinded, Placebo-controlled, Multiple Ascending Dose Phase 1 Clinical Trial to Evaluate Safety, Tolerability, Pharmacokinetics and Pharmacodynamics After Oral Administrations of ID110521156 in Healthy Subjects
Brief Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of ID110521156 in Healthy Adult Subjects
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: IlDong Pharmaceutical Co Ltd (Industry)
Collaborators: YUNOVIA CO.,LTD. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: ID110521156-T2DM-102
Record Dates: First submitted 2024-10-02; First posted 2024-10-10 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Healthy Adult Subjects

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cohort 1 (Experimental): Cohort 1 will consist of 12 healthy subjects, randomly assigned to ID110521156 (10 patients) or its placebo (2 patients)
  Interventions: Drug: ID110521156; Drug: Placebo of 110521156
- Cohort 2 (Experimental): Cohort 2 will consist of 12 healthy subjects, randomly assigned to ID110521156 (10 patients) or its placebo (2 patients)
  Interventions: Drug: ID110521156; Drug: Placebo of 110521156
- Cohort 3 (Experimental): Cohort 3 will consist of 12 healthy subjects, randomly assigned to ID110521156 (10 patients) or its placebo (2 patients)
  Interventions: Drug: ID110521156; Drug: Placebo of 110521156

INTERVENTIONS:
Drug: ID110521156 — ID110521156 capsules taken orally once daily
Drug: Placebo of 110521156 — ID110521156 placebo capsules taken orally once daily

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of multiple oral doses of ID110521156 in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects aged 19 to 50 years at the time of Screening.
* Body mass index (BMI) within ≥27 kg/m2; and a total body weight ≥ 50 kg
* Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study
* For female subjects, not pregnant or lactation women, or naturally menopausal (spontaneous amenorrhea for at least 12 months) or surgically infertility (bilateral tubal occlusion, hysterectomy, bilateral salpingectomy, bilateral oophorectomy etc).

Exclusion Criteria:

* Evidence or history of clinically significant hepatic, renal, neurological, immunological, pulmonary, gastrointestinal (including pancreatitis), endocrine, hematological, cardiovascular, urinary, psychiatric disease, sexual dysfunction or drug allergies.
* Treatment with an investigational drug (including a bioequivalence study) within 180 days prior to the scheduled date of first administration of the investigational product.
* Fertile male subjects who are unwilling or unable to use a highly effective method of contraception for the duration of the study and for at least 90 days after the last dose.

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-11-13 (Actual); Primary Completion 2025-06-19 (Estimated); Study Completion 2025-06-19 (Estimated)

PRIMARY OUTCOMES:
AEs/serious AEs (SAEs) | Throughout study duration, up to 47 days

SECONDARY OUTCOMES:
Maximum concentration of drug in plasma (Cmax) | Day 1 and Day 28
  To assess the PK of ID110521156 when given at single and multiple ascending doses in healthy participants.
Area under the plasma drug concentration-time curve during a dosing interval (AUCtau) | Day 1 and Day 28
  To assess the PK of ID110521156 when given at single and multiple ascending doses in healthy participants.
The time of peak concentration (Tmax) | Day 1 and Day 28
  To assess the PK of ID110521156 when given at single and multiple ascending doses in healthy participants.
Terminal half-life (t1/2) | Day 1 and Day 28
  To assess the PK of ID110521156 when given at single and multiple ascending doses in healthy participants.
Apparent clearance (CL/F) | Day 1 and Day 28
  To assess the PK of ID110521156 when given at single and multiple ascending doses in healthy participants.
Apparent volume of distribution after extravascular administration (Vd/F) | Day 1 and Day 28
  To assess the PK of ID110521156 when given at single and multiple ascending doses in healthy participants.
Renal clearance (CLR) | Day 1 and Day 28
  To assess the PK of ID110521156 when given at single and multiple ascending doses in healthy participants.
fe | Day 1 and Day 28
  To assess the PK of ID110521156 when given at single and multiple ascending doses in healthy participants.
Trough plasma concentration taken directly before the next dose (Ctrough) | Throughout study duration, up to 27 days
  To assess the PK of ID110521156 when given at single and multiple ascending doses in healthy participants.
Minimum concentration of drug in plasma at steady state (Cmin, ss) | Day 28
  To assess the PK of ID110521156 when given at multiple ascending doses in healthy participants.
Average concentration of drug in plasma at steady state (Cavg, ss) | Day 28
  To assess the PK of ID110521156 when given at multiple ascending doses in healthy participants.
peak to trough fluctuation (PTF) | Day 28
  To assess the PK of ID110521156 when given at multiple ascending doses in healthy participants.
accumulation ratio (R) | Day 28
  To assess the PK of ID110521156 when given at multiple ascending doses in healthy participants.
Serum glucose | up to 28 days
  To assess the pharmacodynamics of ID110521156 when given at single and multiple ascending doses in healthy participants.
Insulin | up to 28 days
  To assess the pharmacodynamics of ID110521156 when given at single and multiple ascending doses in healthy participants.
Hemoglobin A1c (HbA1c) | up to 47 days
  To assess the pharmacodynamics of ID110521156 when given at multiple ascending doses in healthy participants.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided